CLINICAL TRIAL: NCT00681590
Title: Safety of Vitamin D Supplementation in the Elderly
Brief Title: Safety of Vitamin D Supplementation in Older Persons
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Silvina Levis, MD, Professor, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20070018
Record Dates: First submitted 2008-05-15; First posted 2008-05-21 (Estimated); Results first posted 2016-03-07 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2016-12

CONDITIONS: Vitamin D Deficiency
Keywords: vitamin D; deficiency; elderly
MeSH Terms: conditions — Vitamin D Deficiency | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): vitamin D (cholecalciferol) 400 IU daily orally - low dose
  Interventions: Dietary Supplement: cholecalciferol (vitamin D)
- 2 (Active Comparator): vitamin D (cholecalciferol) 2000 IU daily orally - high dose
  Interventions: Dietary Supplement: cholecalciferol (vitamin D)

INTERVENTIONS:
Dietary Supplement: cholecalciferol (vitamin D) — 400 IU daily (low dose)
  Arms: 1
Dietary Supplement: cholecalciferol (vitamin D) — 2000 IU daily (high dose)
  Arms: 2

SUMMARY:
This study will evaluate the safety over 6 months of two different doses of vitamin D (cholecalciferol) in men and women age 65 and older. It will also evaluate if supplementation with vitamin D improves physical performance.

DETAILED DESCRIPTION:
120 ambulatory men and women ages 65 to 95 will be enrolled in this study. Each subject will participate in the clinical trial for 6 months.

Parathyroid hormone, vitamin D, and serum and urinary calcium will be measured periodically. Physical performance will be tested at baseline and throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* ambulatory

Exclusion Criteria:

* hypercalcemia
* hypercalciuria > 4 mg/kg body weight/day
* primary, secondary, or tertiary hyperparathyroidism
* renal insufficiency (serum creatinine > 2 mg/dL )
* history of nephrolithiasis
* treatment with vitamin D (ergocalciferol, cholecalciferol, calcitriol)
* treatment with anticonvulsants
* Paget's disease
* severe cardiac, pulmonary, hepatic, renal, or neurological disease
* life expectancy < 1 year
* participation in another trial

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 105 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvina Levis, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

REFERENCES:
- [Background] Lagari V, Gomez-Marin O, Levis S. The role of vitamin D in improving physical performance in the elderly. J Bone Miner Res. 2013 Oct;28(10):2194-201. doi: 10.1002/jbmr.1949. PMID 23553992
- [Result] Lagari VS, Gomez-Marin O, Levis S. Differences in vitamin D3 dosing regimens in a geriatric community-dwelling population. Endocr Pract. 2012 Nov-Dec;18(6):847-54. doi: 10.4158/EP12081.OR. PMID 22784845
- See also: link to Pubmed abstract — http://www.ncbi.nlm.nih.gov/pubmed/23553992

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D 400 IU: participants received one tablet containing cholecalciferol 400 IU daily orally (low dose)
- Vitamin D 2000 IU: participants received one tablet containing cholecalciferol 2000 IU daily orally (high dose)
Period: Overall Study
Arm/Group | Vitamin D 400 IU | Vitamin D 2000 IU
Started | 34 | 71
Completed | 32 | 59
Not Completed | 2 | 12
Not completed — Withdrawal by Subject | 2 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D 400 IU | Vitamin D 2000 IU | Total
Number analyzed (Participants) | 34 | 71 | 105
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (5.9) | 73.9 (6.7) | 73.5 (6.5)
Gender [Count of Participants; unit: Participants]
  Female | 28 | 59 | 87
  Male | 6 | 12 | 18

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Develop Hypercalcemia
Description: calcium serum levels measured at baseline and at the end of the intervention (6-months)
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Vitamin D 400 IU | Vitamin D 2000 IU
Number analyzed (Participants) | 34 | 71
participants | 0 | 2

2. Secondary Outcome: Change From Baseline in Serum 25-hydroxyvitamin D Levels
Time Frame: baseline and 6 months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Vitamin D 400 IU | Vitamin D 2000 IU
Number analyzed (Participants) | 34 | 71
ng/ml | -0.5 (1) | 6.5 (6)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 6 months of the intervention.
Arm/Group | Vitamin D 400 IU | Vitamin D 2000 IU
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/71
Other Adverse Events (participants affected / at risk) | 0/34 | 2/71
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D 400 IU (N=34) | Vitamin D 2000 IU (N=71)
hypercalcemia (Endocrine disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No